CLINICAL TRIAL: NCT06003686
Title: A Spinal Cord Injury (SCI) Stakeholder-vetted Education Module to Mitigate Early Cardioendocrine Health Risks Occurring After Spinal Cord Injuries.
Brief Title: Spinal Cord Injury Model Systems (SCIMS) - Education Module
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gary Farkas, Principal Investigator, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20230202
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries; Obesity; Cardiometabolic Syndrome
MeSH Terms: conditions — Spinal Cord Injuries; Obesity; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paralyzed Veterans of America (PVA) Cardio-Metabolic Disease (CMD) Consumer Guide Group (Experimental): Hard paper copy of as well as an electronic copy of the guide will be provided to subjects and study staff will provide a general review of the contents of the guide with subjects during their education sessions. Participants will be in this group for 6 months.
  Interventions: Behavioral: PVA Consumer Guide
- WebMD Group (Active Comparator): Subjects will be introduced to WebMD and its contents. A brief document will be provided that includes site summary and website. Study staff will provide a very brief overview of the site. Participants will be in this group for 6 months.
  Interventions: Behavioral: WebMD

INTERVENTIONS:
Behavioral: PVA Consumer Guide — Subject's will receive education on the PVA consumer guide 3 times over the course of the study.
  Each session will be approximately 10-15 minutes and will consist of a general review of the nutrition, exercise, and general healthy living guidelines content included.
  Arms: Paralyzed Veterans of America (PVA) Cardio-Metabolic Disease (CMD) Consumer Guide Group
Behavioral: WebMD — Subject's will receive education on how to navigate the WebMD site and find information on health, exercise and nutrition 3 times over the course of the study. Each session will be approximately 10-15 minutes and will consist of a general review of the health and wellness content available on the website. At study completion, subjects in this group will be provided with the PVA guide and a brief orientation of the nutrition, exercise, and general healthy living guidelines content included in the guide.
  Arms: WebMD Group

SUMMARY:
The purpose of this study is to find out if receiving education regarding increased risks of cardiometabolic disease helps subjects understand these risks and how these risks participants' health.

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women with SCI/D aged 18-70 years.
2. Neurologically complete and incomplete American Spinal Injury Association (ASIA) Impairment scale (AIS) A-D spinal cord levels C5 and below.
3. Enrolled no later than 4 months following discharge from initial rehabilitation from SCI.

Exclusion Criteria:

1. Pregnancy determined by urine testing in sexually active females.
2. Cognitive impairment that compromises the legitimacy of consent.
3. Grade 3-4 pressure injury at the time of study entry.
4. Prisoners

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Effectiveness of education modules as determined in the Knowledge Test | baseline, up to 6 months
  Effectiveness as determined by the number of correct answers on the Knowledge Test where the higher number of correct answers indicates increased knowledge of the information provided.

SECONDARY OUTCOMES:
Change in Body Weight as determined by kilograms (kg) | baseline, up to 6 months
  Body weight will be measured in kilograms
Change in Body composition as determined by Dual X-ray Absorptiometry (DXA) | baseline, up to 6 months
  Body composition will be measured in grams using DXA
Change in Body composition as determined by Dual X-ray Absorptiometry (DXA) in Percentage | baseline, up to 6 months
  Body composition will be expressed as a percentage of body fat (BF) using DXA
Change in sugar metabolism as determined by Insulin resistance (IR) | baseline, up to 6 months
  Sugar metabolism will be determined as IR calculated using the formula (fasting serum glucose*fasting serum insulin/22.5). Lower values indicate a higher degree of insulin sensitivity. Fasting values are obtained from blood samples
Change in Quality of Life (QoL) as measured by Quality Index Spinal Cord Injury Version III | baseline, up to 6 months
  A composite score will be obtained to assess change in QoL using a six-point Likert scale. Scores for satisfaction section range from "1- very satisfied" to "6-very dissatisfied". On the important section scoring ranges from "1-very important" to "6- very unimportant"
Change in Quality of Life (QoL) Using the International Spinal Cord Injury Basic Data Set | baseline, up to 6 months
  QoL values will be determined using a scale ranging from 0 (completely dissatisfied) to 10 (completely satisfied).
Change in heart disease risk as determined by cholesterol | baseline, up to 6 months.
  Risk of heart disease will be measured from a blood sample in mg/dL
Change in heart disease risk as determined by blood pressure (BP) | baseline, up to 6 months.
  BP will be measured in mmHg using an arm cuff

CONTACTS AND LOCATIONS:
Overall Officials: Gary Farkas, PhD, Principal Investigator — University of Miami
Locations (3):
- United States (3):
  - MedStar National Rehabilitation Network, Washington D.C., District of Columbia
  - University of Miami - Miami Project to Cure Paralysis, Miami, Florida
  - Baylor Scott & White Institute for Research, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No